CLINICAL TRIAL: NCT04381468
Title: SEMA4D Blockade Safety and Brain Metabolic Activity in Alzheimer's Disease (AD): A Multi-center, Randomized, Double-Blind, Placebo-Controlled Safety and Biomarker Study of Pepinemab Anti-SEMA4D Antibody in Early-AD
Brief Title: SEMA4D Blockade Safety and Brain Metabolic Activity in Alzheimer's Disease (AD)
Acronym: SIGNAL-AD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vaccinex Inc. (Industry)
Collaborators: Alzheimer's Drug Discovery Foundation (Other); Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX15/2503-11
Record Dates: First submitted 2020-05-01; First posted 2020-05-08 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease
Keywords: Mild Cognitive Impairment; Mild Alzheimer's Dementia; Early Alzheimer's Disease; VX15/2503; Semaphorin 4D; SEMA4D; monoclonal antibody
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — pepinemab

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two treatment arms and will receive one dose of study drug every 4 weeks during the 44-week dosing period for a total of 12 doses of study drug
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- pepinemab 40mg/kg (Experimental): The study drug, pepinemab, will be administered via monthly intravenous infusions.
  Interventions: Drug: Pepinemab
- Placebo (Placebo Comparator): .A placebo control will be administered via monthly intravenous infusions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pepinemab — Pepinemab is a humanized IgG4 monoclonal antibody. The antibody is formulated at 20 mg/mL in 20 mM Sodium Acetate buffer, pH 5.4, containing 130 mM Sodium Chloride and 0.02% Polysorbate 80
  Arms: pepinemab 40mg/kg
Drug: Placebo — Placebo consists of formulation buffer only which is 20 mM Sodium Acetate buffer, pH 5.4, containing 130 mM Sodium Chloride and 0.02% Polysorbate 80
  Arms: Placebo

SUMMARY:
To investigate safety, tolerability, the effects on cognition and brain metabolism of pepinemab in early AD dementia (early AD) subjects.

DETAILED DESCRIPTION:
To investigate safety, tolerability, the effects on cognition and brain metabolism of pepinemab, administered as IV infusions every 4 weeks for 44 weeks (12 infusions) in mild dementia due to Alzheimer's Disease (AD)) participants. Participants will be randomized 1:1 to receive 40 mg/kg pepinemab or placebo.

This is a randomized double-blind, placebo-controlled study of pepinemab in mild dementia due to AD. The study is 52 weeks in duration, including a safety and efficacy evaluation 4 weeks after the last dose of study drug. Participants with resolved adverse events at Week 48 will have a safety telephone call at Week 52. Participants with unresolved adverse events at Week 48 will have a safety in-office visit at Week 52. The study protocol will include two sentinel participants in each of the two blinded dose arms. Sentinel dosing will be implemented by randomly assigning one study participant to one of the two dose arms in a blinded manner, treating those participants with study drug. If no unexpected serious adverse events are observed within 48 hours after the first and second participants receive treatment, two additional participants will be enrolled, with one participant assigned randomly to each of the two dose arms. Again a 48-hour safety period will be observed following treatment of the fourth participant to document any unexpected safety events that may occur. Should no unexpected serious adverse events occur within 48 hours after the third and fourth participants receive treatment, the remaining participants will be assigned to the study dose arms according to the blinded randomization scheme and the 1:1 randomization ratio. Participants will be randomized to one of two treatment arms and will receive one dose of study drug every 4 weeks during the 44-week dosing period for a total of 12 doses of study drug. The primary objective is the safety and tolerability of study drug. A key secondary objective is the change in brain metabolism as assessed by [18F]fluorodeoxyglucose (FDG)-PET in the resting state.

ELIGIBILITY:
Inclusion

1. Written informed consent from the participant and legally acceptable representative (trial partner).
2. Have a reliable and competent trial partner who must have a close relationship with the participant, who has face to face contact at least three days a week for a minimum of ten waking hours a week and is willing to accompany the participant to all trial visits. The trial partner should understand the nature of the trial and adhere to trial requirements (e.g., dose, visit schedules, receive phone calls, and evaluations).
3. Male and female participants between the ages of 55 to 85 (inclusive).
4. If female, not be of childbearing potential as indicated by one of the following:

   a. Has reached natural menopause defined as either: i. ≥ 12 months of spontaneous amenorrhea or ii. ≥ 6 months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) levels > 40 mIU/ml as determined by the central laboratory; b. Has had a hysterectomy; or c. Has had a bilateral tubal ligation; or d. Has had a bilateral oophorectomy (with or without a hysterectomy) and more than 6 weeks have passed since the surgery.
5. If male, must agree to use a reliable method of birth control (condoms with contraceptive forms or sexual abstinence) during the study and for 6 months after the last dose of study drug.
6. Must fulfill one of the following:

   1. A documented amyloid PET scan (florbetaben F18, florbetapir F18, or flutametamol F18) determined as positive by the Investigator obtained at any time prior to the Screening visit; or
   2. A documented positive amyloid CSF result obtained at any time prior to the Screening visit; or
   3. Investigator has knowledge of positive amyloid PET scan or positive amyloid CSF result obtained previously; or
   4. A positive amyloid CSF result at screening. The cut-off value for CSF Aβ1-42 or CSF Aβ1-42/Aβ1-40 ratio will be based on the value determined by Vaccinex
7. Evidence of cognitive impairment based on history and neuropsychological testing that meet the diagnostic criteria for probable Alzheimer's dementia.
8. Global Clinical Dementia Rating (CDR) of 0.5 or 1.0
9. MMSE score of 17-26, inclusive.
10. Adequate vision, hearing, and motor function to comply with testing.
11. If receiving medications for AD (including but not limited to donepezil, rivastigmine, galantamine, tacrine, and memantine), be on a stable dose for at least 8 weeks prior to Screening Visit.
12. If on stable doses of centrally-acting medications, be on a stable dose for 8 weeks prior to Screening Visit.
13. In the opinion of the Investigator, is in reasonably good health over the last 6 months and any chronic disease is stable based on medical history and screening assessments.

Exclusion

1. Inability to comply with visit schedule or other protocol requirements.
2. Have participated in an investigational drug or device study within 30 days of the Baseline Visit. If previous investigational drug was a monoclonal antibody, antibody-drug conjugate, or similar protein therapeutic, 180 days or 5 half-lives, whichever occurs first.
3. Have a known allergy to any ingredient in the study drug formulation.
4. Have a body weight greater than 125 kg.
5. Are a suicide risk, as determined by meeting any of the following criteria:

   1. Suicide attempt within one year prior to the Baseline Visit.
   2. Suicidal ideation as defined by a positive response to question 4 and 5 on the C-SSRS within 60 days of the Baseline Visit.
6. Have a history of substance abuse (based on DSMIV criteria) within the past 12 months prior to Screening.
7. Significant acute or chronic infection at Screening including, among others: Known history of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (defined as, HBV surface antigen positive or positive HCV antibody with reflex to positive HCV RNA) at Screening.
8. Have clinically significant laboratory or ECG abnormalities at Screening in the opinion of the Investigator.
9. Have clinically relevant hematologic, hepatic, cardiac, or renal disease.
10. Have a clinically significant medical, surgical, laboratory, or behavioral abnormality which in the judgment of the Investigator makes the participant unsuitable for the study, as well as anyone with a history of malignancy of any type within 2 years of Screening. Persons with a history of surgically excised non-melanoma skin cancers, superficial bladder or prostate cancer are permitted.
11. Participants who have a diagnosis of a neurological condition causing cognitive impairment other than sporadic mild dementia due to AD (e.g., Lewy body disease or frontotemporal dementia), a primary psychiatric diagnosis (e.g., Cognitive Impairment due to Schizophrenia, CIAS), history of frequent concussions or significant findings on brain MRI at screening inconsistent with AD (e.g., cerebrovascular disease or tumor).
12. Have any of the following conditions (which would exclude MRI or PET participation):

    1. Participants deemed unable to cooperate due to claustrophobia, inability to lie on scanner bed for 45 minutes, or inability to achieve venous access sufficient for tracer or pepinemab administration.
    2. An implant/device/condition that is contraindicated for MRI (e.g., pacemaker, severe claustrophobia, prosthetic heart valve, any metal fragments in the eyes or body--in some cases, an X-ray may be needed before an MRI scan, to ensure it is safe to enter the scanner).
    3. Body habitus that would impede completion of imaging scans.
13. Has an MRI scan obtained at Screening that shows evidence of a neurological disorder other than early AD or > 4 cerebral microhemorrhages (regardless of their anatomical location or diagnostic characterization as "possible" or "definite"), a single area of superficial siderosis,
14. Any other clinically significant finding on MRI (e.g., any lesion that may account for their cognitive impairment, including but not limited to brain tumor, severe white matter disease arteriovenous malformation, cavernous hemangioma, or any infarct in a strategic cortical or subcortical location).
15. Are undergoing FDG-PET and have received research-related radiation exposure that exceeds institutional guidelines in the prior year if applicable.
16. Are undergoing a LP for CSF collection and have any of the following conditions: uncorrected bleeding or clotting disorders, skin infections near the site of the LP, suspicion of increased intracranial pressure, allergies to numbing medications (local anesthetics), acute spinal trauma.
17. Are undergoing a LP for CSF collection and taking any of the following types of anticoagulants: coumarins and indandiones, Factor Xa inhibitors, heparins, or thrombin inhibitors.
18. Has received treatment with any FDA accelerated approval therapy for treatment of Alzheimer's Disease
19. Has a Screening MRI that shows Amyloid-related imaging abnormalities edema (ARIA-E)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment emergent adverse events (TEAEs) | Up to 40 weeks
  TEAEs are defined as Adverse events (AEs) with onset after date-time of first dose, or medical conditions present prior to the start of IP but increased in severity or relationship after date-time of first dose of IP.

SECONDARY OUTCOMES:
Effects on brain metabolism | Up to 36 weeks
  As assessed by [18F]fluorodeoxyglucose (FDG)-PET in the resting state following administration of 20 mg/kg or 40 mg/kg pepinemab or placebo.
Alzheimer's Disease Assessment Scale- Cognitive subscale (ADAS-cog13) | Up to 36 weeks
  The Alzheimer's Disease Assessment Scale (ADAS-cog13) will be performed to test the cognition of subjects. The score ranges from 0 to 75，and higher values represent a better outcome.
Clinical Dementia Rating (CDR) | Up to 36 weeks
  The CDR assesses 3 domains of cognition (memory, orientation, judgment/problem solving) and 3 domains of function (community affairs, home/hobbies, personal care) using semi-structured interviews of both the study subject and an informant carried out by a trained rater. The CDR is scored using a standard methodology. Each domain is rated on a 5-point scale and lower numbers represent a better outcome.
Mini Mental State Examination (MMSE) | Up to 36 weeks
  Mini-Mental State Examination scores(MMSE) will be performed to test the cognition of subjects. The score ranges from 0 to 30，and higher values represent a better outcome.
Alzheimer's Disease Cooperative Study - Activities of Daily Living | Up to 36 weeks
  The ADCS-ADL assesses the competence of participants with AD in basic and instrumental activities of daily living (ADLs). It is administered by a clinician as a structured interview with a caregiver. The maximum score is 30. A higher score is better.
Alzheimer's Disease Cooperative Study- Clinical Global Impression of Change (ADCS-CGIC) | Up to 36 weeks
  The ADCS-CGIC focuses on clinicians' observations of change in the patient's cognitive, functional, and behavioral performance since the beginning of a trial. The ADCS-CGIC gives a discrete score that ranges from 1-7 with 7 being the worst outcome.
Neuropsychiatric Inventory (NPI) | Up to 36 weeks
  The NPI is a trial partner interview-based rating scale assessing 12 behavioral disturbances occurring in dementia subjects. Items are scored for both frequency and severity. Total scores range from 0-144 with higher scores indicating greater behavioral disturbances. For each item, the associated trial partner distress is also assessed.
Immunogenicity of pepinemab in serum | Up to 36 weeks
  As assessed by the frequency and titer of anti-drug antibodies.

OTHER OUTCOMES:
Peak serum concentration (Cmax) | Up to 36 weeks
  PK parameter
Area under the serum concentration vs. time curve (AUC) | Up to 36 weeks
  PK parameter
Half-life of pepinemab | Up to 36 weeks
  PK parameter
Serum and CSF levels of neuroinflammatory cytokines | Up to 36 weeks
  IL-1, IL-2, IL-4, IL-5, IL-6, IL-10, IL-12, IL13,IFNγ, TNF-α, TGFβ
T- and B-Cell Quantitation by Flow Cytometry (TBNK) | Up to 36 weeks
  B cells, total count; Natural killer (NK) cells, total count; T cells, total count; Absolute CD4/CD8 count with ratio
Plasma and CSF concentration of neurofilament light chain (NfL) | Up to 36 weeks
Plasma and CSF concentrations of Aβ1-42/Aβ1-40 | Up to 36 weeks
CSF levels of pepinemab | Up to 36 weeks
CSF concentrations of tau and p-tau | Up to 36 weeks
CSF concentrations of YKL-40 | Up to 36 weeks
Cellular SEMA4D levels | Up to 36 weeks
  PD parameter to determine the level of SEMA4D expression on T lymphocytes
Total soluble SEMA4D levels | Up to 36 weeks
  PD parameter to determine levels of total soluble SEMA4D
Effects on brain volume | Up to 36 weeks
  As measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Eric Siemers, MD, Study Director — Vaccinex Inc.
Locations (14):
- United States (14):
  - Pacific Research Network, Inc, San Diego, California
  - Georgetown University, Washington D.C., District of Columbia
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - JEM Research Institute, Lake Worth, Florida
  - Premiere Research Institute of Palm Beach, Neurology, Palm Beach, Florida
  - Brain Matters Research, Stuart, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center, Fairway, Kansas
  - Neurological Associates of Albany, Albany, New York
  - Dent Neurological Associates, Amherst, New York
  - Columbia University Irving Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Re-Cognition Health, Fairfax, Virginia

REFERENCES:
- [Background] Hardy JA, Higgins GA. Alzheimer's disease: the amyloid cascade hypothesis. Science. 1992 Apr 10;256(5054):184-5. doi: 10.1126/science.1566067. No abstract available.
- [Background] Selkoe DJ. Resolving controversies on the path to Alzheimer's therapeutics. Nat Med. 2011 Sep 7;17(9):1060-5. doi: 10.1038/nm.2460. PMID 21900936
- [Background] Moreau-Fauvarque C, Kumanogoh A, Camand E, Jaillard C, Barbin G, Boquet I, Love C, Jones EY, Kikutani H, Lubetzki C, Dusart I, Chedotal A. The transmembrane semaphorin Sema4D/CD100, an inhibitor of axonal growth, is expressed on oligodendrocytes and upregulated after CNS lesion. J Neurosci. 2003 Oct 8;23(27):9229-39. doi: 10.1523/JNEUROSCI.23-27-09229.2003. PMID 14534257
- [Background] Fisher, T. L., J. E. Leonard, and E. Smith. 2019. Investigator's Brochure : pepinemab-Neurology. Version 4 ed. Vaccinex, Inc.
- [Background] Basile JR, Gavard J, Gutkind JS. Plexin-B1 utilizes RhoA and Rho kinase to promote the integrin-dependent activation of Akt and ERK and endothelial cell motility. J Biol Chem. 2007 Nov 30;282(48):34888-95. doi: 10.1074/jbc.M705467200. Epub 2007 Sep 12. PMID 17855350
- [Background] Giraudon P, Vincent P, Vuaillat C, Verlaeten O, Cartier L, Marie-Cardine A, Mutin M, Bensussan A, Belin MF, Boumsell L. Semaphorin CD100 from activated T lymphocytes induces process extension collapse in oligodendrocytes and death of immature neural cells. J Immunol. 2004 Jan 15;172(2):1246-55. doi: 10.4049/jimmunol.172.2.1246. PMID 14707103
- [Background] Giraudon P, Vincent P, Vuaillat C. T-cells in neuronal injury and repair: semaphorins and related T-cell signals. Neuromolecular Med. 2005;7(3):207-16. doi: 10.1385/NMM:7:3:207. PMID 16247181
- [Background] Okuno T, Nakatsuji Y, Moriya M, Takamatsu H, Nojima S, Takegahara N, Toyofuku T, Nakagawa Y, Kang S, Friedel RH, Sakoda S, Kikutani H, Kumanogoh A. Roles of Sema4D-plexin-B1 interactions in the central nervous system for pathogenesis of experimental autoimmune encephalomyelitis. J Immunol. 2010 Feb 1;184(3):1499-506. doi: 10.4049/jimmunol.0903302. Epub 2009 Dec 28. PMID 20038643
- [Background] Smith ES, Jonason A, Reilly C, Veeraraghavan J, Fisher T, Doherty M, Klimatcheva E, Mallow C, Cornelius C, Leonard JE, Marchi N, Janigro D, Argaw AT, Pham T, Seils J, Bussler H, Torno S, Kirk R, Howell A, Evans EE, Paris M, Bowers WJ, John G, Zauderer M. SEMA4D compromises blood-brain barrier, activates microglia, and inhibits remyelination in neurodegenerative disease. Neurobiol Dis. 2015 Jan;73:254-68. doi: 10.1016/j.nbd.2014.10.008. Epub 2014 Oct 18. PMID 25461192
- [Background] Van Raamsdonk JM, Gibson WT, Pearson J, Murphy Z, Lu G, Leavitt BR, Hayden MR. Body weight is modulated by levels of full-length huntingtin. Hum Mol Genet. 2006 May 1;15(9):1513-23. doi: 10.1093/hmg/ddl072. Epub 2006 Mar 28. PMID 16571604
- [Background] Van Raamsdonk JM, Murphy Z, Slow EJ, Leavitt BR, Hayden MR. Selective degeneration and nuclear localization of mutant huntingtin in the YAC128 mouse model of Huntington disease. Hum Mol Genet. 2005 Dec 15;14(24):3823-35. doi: 10.1093/hmg/ddi407. Epub 2005 Nov 8. PMID 16278236
- [Background] Carroll JB, Lerch JP, Franciosi S, Spreeuw A, Bissada N, Henkelman RM, Hayden MR. Natural history of disease in the YAC128 mouse reveals a discrete signature of pathology in Huntington disease. Neurobiol Dis. 2011 Jul;43(1):257-65. doi: 10.1016/j.nbd.2011.03.018. Epub 2011 Mar 31. PMID 21458571
- [Background] Southwell AL, Franciosi S, Villanueva EB, Xie Y, Winter LA, Veeraraghavan J, Jonason A, Felczak B, Zhang W, Kovalik V, Waltl S, Hall G, Pouladi MA, Smith ES, Bowers WJ, Zauderer M, Hayden MR. Anti-semaphorin 4D immunotherapy ameliorates neuropathology and some cognitive impairment in the YAC128 mouse model of Huntington disease. Neurobiol Dis. 2015 Apr;76:46-56. doi: 10.1016/j.nbd.2015.01.002. Epub 2015 Feb 3. PMID 25662335
- [Background] Patnaik A, Weiss GJ, Leonard JE, Rasco DW, Sachdev JC, Fisher TL, Winter LA, Reilly C, Parker RB, Mutz D, Blaydorn L, Tolcher AW, Zauderer M, Ramanathan RK. Safety, Pharmacokinetics, and Pharmacodynamics of a Humanized Anti-Semaphorin 4D Antibody, in a First-In-Human Study of Patients with Advanced Solid Tumors. Clin Cancer Res. 2016 Feb 15;22(4):827-36. doi: 10.1158/1078-0432.CCR-15-0431. Epub 2015 Oct 7. PMID 26446947
- [Background] LaGanke C, Samkoff L, Edwards K, Jung Henson L, Repovic P, Lynch S, Stone L, Mattson D, Galluzzi A, Fisher TL, Reilly C, Winter LA, Leonard JE, Zauderer M. Safety/tolerability of the anti-semaphorin 4D Antibody VX15/2503 in a randomized phase 1 trial. Neurol Neuroimmunol Neuroinflamm. 2017 Jun 16;4(4):e367. doi: 10.1212/NXI.0000000000000367. eCollection 2017 Jul. PMID 28642891
- [Background] Verkhratsky A, Zorec R, Parpura V. Stratification of astrocytes in healthy and diseased brain. Brain Pathol. 2017 Sep;27(5):629-644. doi: 10.1111/bpa.12537. PMID 28805002
- [Background] Tremblay ME, Stevens B, Sierra A, Wake H, Bessis A, Nimmerjahn A. The role of microglia in the healthy brain. J Neurosci. 2011 Nov 9;31(45):16064-9. doi: 10.1523/JNEUROSCI.4158-11.2011. PMID 22072657
- [Background] Saab AS, Tzvetavona ID, Trevisiol A, Baltan S, Dibaj P, Kusch K, Mobius W, Goetze B, Jahn HM, Huang W, Steffens H, Schomburg ED, Perez-Samartin A, Perez-Cerda F, Bakhtiari D, Matute C, Lowel S, Griesinger C, Hirrlinger J, Kirchhoff F, Nave KA. Oligodendroglial NMDA Receptors Regulate Glucose Import and Axonal Energy Metabolism. Neuron. 2016 Jul 6;91(1):119-32. doi: 10.1016/j.neuron.2016.05.016. Epub 2016 Jun 9. PMID 27292539
- [Background] Boillee S, Yamanaka K, Lobsiger CS, Copeland NG, Jenkins NA, Kassiotis G, Kollias G, Cleveland DW. Onset and progression in inherited ALS determined by motor neurons and microglia. Science. 2006 Jun 2;312(5778):1389-92. doi: 10.1126/science.1123511. PMID 16741123
- [Background] Yamanaka K, Chun SJ, Boillee S, Fujimori-Tonou N, Yamashita H, Gutmann DH, Takahashi R, Misawa H, Cleveland DW. Astrocytes as determinants of disease progression in inherited amyotrophic lateral sclerosis. Nat Neurosci. 2008 Mar;11(3):251-3. doi: 10.1038/nn2047. Epub 2008 Feb 3. PMID 18246065
- [Background] Benraiss A, Wang S, Herrlinger S, Li X, Chandler-Militello D, Mauceri J, Burm HB, Toner M, Osipovitch M, Jim Xu Q, Ding F, Wang F, Kang N, Kang J, Curtin PC, Brunner D, Windrem MS, Munoz-Sanjuan I, Nedergaard M, Goldman SA. Human glia can both induce and rescue aspects of disease phenotype in Huntington disease. Nat Commun. 2016 Jun 7;7:11758. doi: 10.1038/ncomms11758. PMID 27273432
- [Background] Heneka MT, Carson MJ, El Khoury J, Landreth GE, Brosseron F, Feinstein DL, Jacobs AH, Wyss-Coray T, Vitorica J, Ransohoff RM, Herrup K, Frautschy SA, Finsen B, Brown GC, Verkhratsky A, Yamanaka K, Koistinaho J, Latz E, Halle A, Petzold GC, Town T, Morgan D, Shinohara ML, Perry VH, Holmes C, Bazan NG, Brooks DJ, Hunot S, Joseph B, Deigendesch N, Garaschuk O, Boddeke E, Dinarello CA, Breitner JC, Cole GM, Golenbock DT, Kummer MP. Neuroinflammation in Alzheimer's disease. Lancet Neurol. 2015 Apr;14(4):388-405. doi: 10.1016/S1474-4422(15)70016-5. PMID 25792098
- [Background] Gonzalez-Reyes RE, Nava-Mesa MO, Vargas-Sanchez K, Ariza-Salamanca D, Mora-Munoz L. Involvement of Astrocytes in Alzheimer's Disease from a Neuroinflammatory and Oxidative Stress Perspective. Front Mol Neurosci. 2017 Dec 19;10:427. doi: 10.3389/fnmol.2017.00427. eCollection 2017. PMID 29311817
- [Background] Jonsson T, Stefansson H, Steinberg S, Jonsdottir I, Jonsson PV, Snaedal J, Bjornsson S, Huttenlocher J, Levey AI, Lah JJ, Rujescu D, Hampel H, Giegling I, Andreassen OA, Engedal K, Ulstein I, Djurovic S, Ibrahim-Verbaas C, Hofman A, Ikram MA, van Duijn CM, Thorsteinsdottir U, Kong A, Stefansson K. Variant of TREM2 associated with the risk of Alzheimer's disease. N Engl J Med. 2013 Jan 10;368(2):107-16. doi: 10.1056/NEJMoa1211103. Epub 2012 Nov 14. PMID 23150908
- [Background] Walter J. The Triggering Receptor Expressed on Myeloid Cells 2: A Molecular Link of Neuroinflammation and Neurodegenerative Diseases. J Biol Chem. 2016 Feb 26;291(9):4334-41. doi: 10.1074/jbc.R115.704981. Epub 2015 Dec 22. PMID 26694609
- [Background] Hong S, Beja-Glasser VF, Nfonoyim BM, Frouin A, Li S, Ramakrishnan S, Merry KM, Shi Q, Rosenthal A, Barres BA, Lemere CA, Selkoe DJ, Stevens B. Complement and microglia mediate early synapse loss in Alzheimer mouse models. Science. 2016 May 6;352(6286):712-716. doi: 10.1126/science.aad8373. Epub 2016 Mar 31. PMID 27033548
- [Background] Halassa MM, Fellin T, Haydon PG. The tripartite synapse: roles for gliotransmission in health and disease. Trends Mol Med. 2007 Feb;13(2):54-63. doi: 10.1016/j.molmed.2006.12.005. Epub 2007 Jan 4. PMID 17207662
- [Background] Barres BA. The mystery and magic of glia: a perspective on their roles in health and disease. Neuron. 2008 Nov 6;60(3):430-40. doi: 10.1016/j.neuron.2008.10.013. PMID 18995817
- [Background] Fisher TL, Reilly CA, Winter LA, Pandina T, Jonason A, Scrivens M, Balch L, Bussler H, Torno S, Seils J, Mueller L, Huang H, Klimatcheva E, Howell A, Kirk R, Evans E, Paris M, Leonard JE, Smith ES, Zauderer M. Generation and preclinical characterization of an antibody specific for SEMA4D. MAbs. 2016;8(1):150-62. doi: 10.1080/19420862.2015.1102813. Epub 2015 Oct 2. PMID 26431358
- [Background] Cai Z, Qiao PF, Wan CQ, Cai M, Zhou NK, Li Q. Role of Blood-Brain Barrier in Alzheimer's Disease. J Alzheimers Dis. 2018;63(4):1223-1234. doi: 10.3233/JAD-180098. PMID 29782323
- [Background] Reiman EM, Jagust WJ. Brain imaging in the study of Alzheimer's disease. Neuroimage. 2012 Jun;61(2):505-16. doi: 10.1016/j.neuroimage.2011.11.075. Epub 2011 Dec 7. PMID 22173295
- [Background] Lange C, Suppa P, Frings L, Brenner W, Spies L, Buchert R. Optimization of Statistical Single Subject Analysis of Brain FDG PET for the Prognosis of Mild Cognitive Impairment-to-Alzheimer's Disease Conversion. J Alzheimers Dis. 2016;49(4):945-959. doi: 10.3233/JAD-150814. PMID 26577523